CLINICAL TRIAL: NCT07086469
Title: A Prospective, Single-arm, Phase II Clinical Trial of Surufatinib in Combination With Neoadjuvant Chemo-immunotherapy and Concurrent Chemoradiotherapy for Patients With Unresectable Locally Advanced Esophageal Squamous Cell Carcinoma
Brief Title: Surufatinib in Combination With Neoadjuvant Chemo-immunotherapy and Concurrent Chemoradiotherapy for Patients With Unresectable Locally Advanced Esophageal Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Liu, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GASTO-10132
Record Dates: First submitted 2025-07-15; First posted 2025-07-25 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Toripalimab; Surufatinib; Neoadjuvant Immunochemotherapy; Chemoradiotherapy; Esophageal Squamous Cell Carcinoma
Keywords: Toripalimab; Surufatinib; Neoadjuvant Immunochemotherapy; Chemoradiotherapy; Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The study group (Experimental): Patients will first receive two cycles of neoadjuvant therapy consisting of albumin-bound paclitaxel, cisplatin, toripalimab, and surufatinib. This will be followed by definitive concurrent radiotherapy combined with albumin-bound paclitaxel, cisplatin, toripalimab, and surufatinib.
  Interventions: Drug: Neoadjuvant immunochemotherapy; Drug: Surufatinib Administration; Drug: Concurrent Chemotherapy; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Neoadjuvant immunochemotherapy — Albumin-bound paclitaxel 260 mg/m² on day 1, cisplatin 25 mg/m² on days 1-3, and toripalimab 240 mg on day 1 of each 3-week cycle (q3w), for a total of 2 cycles.
Drug: Surufatinib Administration — Surufatinib 200 mg orally once daily (po, qd) on days 1-14, administered concurrently with immunochemotherapy. During radiotherapy, surufatinib will be administered at the start of each radiotherapy phase.
Drug: Concurrent Chemotherapy — Toripalimab 240 mg on day 1 of each 3-week cycle (q3w), starting one day prior to the initiation of radiotherapy. Weekly administration of albumin-bound paclitaxel 50 mg/m² and cisplatin 25 mg/m² on day 1 during the radiotherapy course.
Radiation: Radiotherapy — All patients will undergo thoracic intensity-modulated radiotherapy (IMRT), delivered once daily, 5 days per week, at a total prescribed dose of 50 Gy.

SUMMARY:
The combination of surufatinib with neoadjuvant chemo-immunotherapy and definitive concurrent chemoradiotherapy represents a promising new therapeutic strategy that may further improve the prognosis of patients with unresectable locally advanced esophageal squamous cell carcinoma (ESCC). Therefore, we propose to conduct a prospective, single-arm, phase II clinical trial to evaluate the efficacy and safety of this regimen in patients with unresectable, locally advanced ESCC.

DETAILED DESCRIPTION:
This is a prospective, single-arm, phase II clinical trial designed to evaluate the efficacy and safety of surufatinib in combination with neoadjuvant chemo-immunotherapy and concurrent chemoradiotherapy in patients with unresectable locally advanced esophageal squamous cell carcinoma. Patients will first receive two cycles of neoadjuvant therapy consisting of albumin-bound paclitaxel, cisplatin, toripalimab, and surufatinib. This will be followed by definitive concurrent chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of esophageal squamous cell carcinoma (ESCC).
* Locally advanced, unresectable esophageal cancer assessed by endoscopic ultrasound and imaging studies, including esophagography, contrast-enhanced CT scans of the lower neck, chest, and upper abdomen, MRI of the lower neck and chest, whole-body bone scintigraphy, or PET/CT; staged as T2-4, N0-3, M0-1 (M1 limited to supraclavicular lymph node metastasis).
* Male or female patients aged 18 to 80 years.
* No prior chemotherapy, radiotherapy, surgery, targeted therapy, or immunotherapy.
* Expected life expectancy of at least 12 weeks.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate organ and bone marrow function defined as: Forced expiratory volume in one second (FEV1) ≥ 1000 mL; Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L; Platelet count ≥ 100 × 10⁹/L; Hemoglobin ≥ 90 g/L; Creatinine clearance ≥ 50 mL/min calculated by the Cockcroft-Gault formula (Cockcroft and Gault, 1976); Total bilirubin ≤ 1.5 × upper limit of normal (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN.
* Signed and dated informed consent form must be obtained prior to any study-related procedures.

Exclusion Criteria:

* Participation in another clinical trial simultaneously, except for observational (non-interventional) studies.
* Prior use of any targeted therapy.
* Major surgery within 4 weeks prior to study entry (excluding vascular access procedures).
* Uncontrolled comorbidities, including but not limited to active or ongoing infections, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina, arrhythmias, active peptic ulcer disease or gastritis, intestinal perforation, bowel obstruction, active bleeding disorders, or psychiatric/social conditions that may impair compliance with study requirements or the ability to provide informed consent.
* Performance status (PS) score of 2-4.
* Presence of any of the following organ or bone marrow dysfunctions: Forced expiratory volume in one second (FEV1) < 1000 mL; Absolute neutrophil count (ANC) < 1.5 × 10⁹/L; Platelet count < 100 × 10⁹/L; Hemoglobin < 90 g/L; Creatinine clearance < 50 mL/min calculated by the Cockcroft-Gault formula (Cockcroft and Gault, 1976); Total bilirubin > 1.5 × upper limit of normal (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) > 2.5 × ULN.
* Any condition that may interfere with the assessment of efficacy or safety of surufatinib.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2025-07-20 (Actual); Primary Completion 2029-07-19 (Estimated); Study Completion 2029-07-19 (Estimated)

PRIMARY OUTCOMES:
2-year progression-free survival rate | 2 years
  The 2-year progression-free survival rate refers to the proportion of patients who remain alive without evidence of disease progression at 24 months after initiation of treatment.

SECONDARY OUTCOMES:
Median overall survival (OS) | 2 years
  The time from the start of treatment to death from any cause.
Objective Response Rate (ORR) | 2 months after CCRT
  The objective response rate refers to the proportion of patients with a measurable reduction in tumor burden, including complete response (CR) and partial response (PR), as defined by standardized criteria such as RECIST (Response Evaluation Criteria in Solid Tumors).
Locoregional Progression-Free Survival (LRPFS) | 2 years
  LRPFS is defined as the time from the start of treatment to the first occurrence of locoregional disease progression or death from any cause.
Distant Metastasis-Free Survival (DMFS) | 2 years
  DMFS refers to the time from treatment initiation to the first occurrence of distant metastasis or death from any cause. It reflects the effectiveness of systemic disease control.
Treatment-related adverse events | 1 year after treatment
  The assessment of treatment-related adverse events (AEs), including their type, severity, frequency, and impact on patients.
Patient-reported quality of life | 1 year after treatment
  Quality of life assessed using the EORTC Quality of Life Core Questionnaire (QLQ-C30).
Patient-reported esophageal-specific symptoms | 1 year after treatment
  Esophageal-specific symptoms assessed using EORTC QLQ-OES18 questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Liu, Principal Investigator — Sun yat-sen universtiy cancer center
Locations (1):
- Sun yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Zhang P, Chen Z, Shi S, Li Z, Ye F, Song L, Zhang Y, Yin F, Zhang X, Xu J, Cheng Y, Su W, Shi M, Fan S, Tan P, Zhong C, Lu M, Shen L. Efficacy and safety of surufatinib plus toripalimab, a chemotherapy-free regimen, in patients with advanced gastric/gastroesophageal junction adenocarcinoma, esophageal squamous cell carcinoma, or biliary tract cancer. Cancer Immunol Immunother. 2024 May 7;73(7):119. doi: 10.1007/s00262-024-03677-7. PMID 38713205
- [Background] Xu J, Shen L, Zhou Z, Li J, Bai C, Chi Y, Li Z, Xu N, Li E, Liu T, Bai Y, Yuan Y, Li X, Wang X, Chen J, Ying J, Yu X, Qin S, Yuan X, Zhang T, Deng Y, Xiu D, Cheng Y, Tao M, Jia R, Wang W, Li J, Fan S, Peng M, Su W. Surufatinib in advanced extrapancreatic neuroendocrine tumours (SANET-ep): a randomised, double-blind, placebo-controlled, phase 3 study. Lancet Oncol. 2020 Nov;21(11):1500-1512. doi: 10.1016/S1470-2045(20)30496-4. Epub 2020 Sep 20. PMID 32966811
- [Background] Xu J, Shen L, Bai C, Wang W, Li J, Yu X, Li Z, Li E, Yuan X, Chi Y, Yin Y, Lou W, Xu N, Bai Y, Zhang T, Xiu D, Wang X, Yuan Y, Chen J, Qin S, Jia R, Lu M, Cheng Y, Zhou Z, Li J, He J, Su W. Surufatinib in advanced pancreatic neuroendocrine tumours (SANET-p): a randomised, double-blind, placebo-controlled, phase 3 study. Lancet Oncol. 2020 Nov;21(11):1489-1499. doi: 10.1016/S1470-2045(20)30493-9. Epub 2020 Sep 20. PMID 32966810
- [Background] Syed YY. Surufatinib: First Approval. Drugs. 2021 Apr;81(6):727-732. doi: 10.1007/s40265-021-01489-y. PMID 33788183
- [Background] Wang J, Yu JP, Wang JL, Ni XC, Sun ZQ, Sun W, Nie B, Jiang JT, Sun SP, Wu CP. [Pathologic response and changes of serum VEGF during chemoradiotherapy may predict prognosis in non-surgical patients with esophageal carcinoma]. Zhonghua Zhong Liu Za Zhi. 2016 Aug;38(8):589-95. doi: 10.3760/cma.j.issn.0253-3766.2016.08.005. Chinese. PMID 27531478
- [Background] Zhu Y, Wen J, Li Q, Chen B, Zhao L, Liu S, Yang Y, Wang S, Lv Y, Li J, Zhang L, Hu Y, Liu M, Xi M. Toripalimab combined with definitive chemoradiotherapy in locally advanced oesophageal squamous cell carcinoma (EC-CRT-001): a single-arm, phase 2 trial. Lancet Oncol. 2023 Apr;24(4):371-382. doi: 10.1016/S1470-2045(23)00060-8. PMID 36990609
- [Background] Shinoda M, Ando N, Kato K, Ishikura S, Kato H, Tsubosa Y, Minashi K, Okabe H, Kimura Y, Kawano T, Kosugi S, Toh Y, Nakamura K, Fukuda H; Japan Clinical Oncology Group. Randomized study of low-dose versus standard-dose chemoradiotherapy for unresectable esophageal squamous cell carcinoma (JCOG0303). Cancer Sci. 2015 Apr;106(4):407-12. doi: 10.1111/cas.12622. Epub 2015 Mar 9. PMID 25640628
- [Background] Suntharalingam M, Winter K, Ilson D, Dicker AP, Kachnic L, Konski A, Chakravarthy AB, Anker CJ, Thakrar H, Horiba N, Dubey A, Greenberger JS, Raben A, Giguere J, Roof K, Videtic G, Pollock J, Safran H, Crane CH. Effect of the Addition of Cetuximab to Paclitaxel, Cisplatin, and Radiation Therapy for Patients With Esophageal Cancer: The NRG Oncology RTOG 0436 Phase 3 Randomized Clinical Trial. JAMA Oncol. 2017 Nov 1;3(11):1520-1528. doi: 10.1001/jamaoncol.2017.1598. PMID 28687830
- [Background] Hulshof MCCM, Geijsen ED, Rozema T, Oppedijk V, Buijsen J, Neelis KJ, Nuyttens JJME, van der Sangen MJC, Jeene PM, Reinders JG, van Berge Henegouwen MI, Thano A, van Hooft JE, van Laarhoven HWM, van der Gaast A. Randomized Study on Dose Escalation in Definitive Chemoradiation for Patients With Locally Advanced Esophageal Cancer (ARTDECO Study). J Clin Oncol. 2021 Sep 1;39(25):2816-2824. doi: 10.1200/JCO.20.03697. Epub 2021 Jun 8. PMID 34101496
- [Background] Conroy T, Galais MP, Raoul JL, Bouche O, Gourgou-Bourgade S, Douillard JY, Etienne PL, Boige V, Martel-Lafay I, Michel P, Llacer-Moscardo C, Francois E, Crehange G, Abdelghani MB, Juzyna B, Bedenne L, Adenis A; Federation Francophone de Cancerologie Digestive and UNICANCER-GI Group. Definitive chemoradiotherapy with FOLFOX versus fluorouracil and cisplatin in patients with oesophageal cancer (PRODIGE5/ACCORD17): final results of a randomised, phase 2/3 trial. Lancet Oncol. 2014 Mar;15(3):305-14. doi: 10.1016/S1470-2045(14)70028-2. Epub 2014 Feb 18. PMID 24556041
- [Background] Xu Y, Dong B, Zhu W, Li J, Huang R, Sun Z, Yang X, Liu L, He H, Liao Z, Guan N, Kong Y, Wang W, Chen J, He H, Qiu G, Zeng M, Pu J, Hu W, Bao Y, Liu Z, Ma J, Jiang H, Du X, Hu J, Zhuang T, Cai J, Huang J, Tao H, Liu Y, Liang X, Zhou J, Tao G, Zheng X, Chen M. A Phase III Multicenter Randomized Clinical Trial of 60 Gy versus 50 Gy Radiation Dose in Concurrent Chemoradiotherapy for Inoperable Esophageal Squamous Cell Carcinoma. Clin Cancer Res. 2022 May 2;28(9):1792-1799. doi: 10.1158/1078-0432.CCR-21-3843. PMID 35190815
- [Background] Minsky BD, Pajak TF, Ginsberg RJ, Pisansky TM, Martenson J, Komaki R, Okawara G, Rosenthal SA, Kelsen DP. INT 0123 (Radiation Therapy Oncology Group 94-05) phase III trial of combined-modality therapy for esophageal cancer: high-dose versus standard-dose radiation therapy. J Clin Oncol. 2002 Mar 1;20(5):1167-74. doi: 10.1200/JCO.2002.20.5.1167. PMID 11870157
- [Background] Cooper JS, Guo MD, Herskovic A, Macdonald JS, Martenson JA Jr, Al-Sarraf M, Byhardt R, Russell AH, Beitler JJ, Spencer S, Asbell SO, Graham MV, Leichman LL. Chemoradiotherapy of locally advanced esophageal cancer: long-term follow-up of a prospective randomized trial (RTOG 85-01). Radiation Therapy Oncology Group. JAMA. 1999 May 5;281(17):1623-7. doi: 10.1001/jama.281.17.1623. PMID 10235156
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338